CLINICAL TRIAL: NCT00436930
Title: Randomized Phase II Trial of Autologous Vaccines Consisting of Adjuvant GM-CSF Plus Proliferating Tumor Cells Versus GM-CSF Plus Dendritic Cells Loaded With Proliferating Tumor Cells in Patients With Metastatic Melanoma (MAC-VAC)
Brief Title: Vaccine Therapy and GM-CSF in Treating Patients With Recurrent or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Robert O. Dillman, Hoag Cancer Institute at Hoag Memorial Hospital Presbyterian
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000530026; HOAG-HCC-06-03
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-06

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — FANG vaccine; sargramostim

ARMS (2):
- Arm I (Experimental): Patients receive irradiated autologous tumor cells subcutaneously (SC) and sargramostim (GM-CSF) SC once weekly for 3 weeks and then once monthly for up to 5 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: autologous tumor cell vaccine; Biological: sargramostim
- Arm II (Experimental): Patients receive autologous dendritic cells loaded with irradiated autologous tumor cells SC and GM-CSF SC once weekly for 3 weeks and then once monthly for up to 5 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: sargramostim; Biological: therapeutic autologous dendritic cells

INTERVENTIONS:
Biological: autologous tumor cell vaccine — Given subcutaneously
  Arms: Arm I
Biological: sargramostim — Given subcutaneously
Biological: therapeutic autologous dendritic cells — Given subcutaneously
  Arms: Arm II

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells. Colony-stimulating factors, such as GM-CSF, increase the number of white blood cells and platelets found in bone marrow or peripheral blood. Giving vaccine therapy together with GM-CSF may be an effective treatment for melanoma.

PURPOSE: This randomized phase II trial is studying two different vaccine therapy regimens to compare how well they work when given together with GM-CSF in treating patients with recurrent or metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival, progression-free survival, event-free survival, and failure-free survival of patients with metastatic melanoma treated with vaccine therapy comprising irradiated autologous tumor cells vs autologous dendritic cells loaded with irradiated autologous tumor cells in combination with sargramostim (GM-CSF).
* Compare the frequency of immune response based on delayed-type hypersensitivity to irradiated autologous tumor cells and serologic and cellular assays at baseline and during and after completion of autologous tumor cell-based vaccine therapy in these patients.
* Compare the safety of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to measurable disease (yes vs no) and location of disease (distant vs regional). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive irradiated autologous tumor cells subcutaneously (SC) and sargramostim (GM-CSF) SC once weekly for 3 weeks and then once monthly for up to 5 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive autologous dendritic cells loaded with irradiated autologous tumor cells SC and GM-CSF SC once weekly for 3 weeks and then once monthly for up to 5 months in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * Regionally recurrent or distant metastatic disease
* Must have an established continuously proliferating cell line expanded to about 200 million cells that is free of stromal cells and contamination
* No active CNS metastases

  * Prior treatment for brain metastases or spinal cord compression allowed
  * No clear evidence of disease progression in the CNS
  * No concurrent pharmacologic doses of corticosteroids

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 70-100% OR ECOG PS 0-1
* Platelet count > 100,000/mm³
* Hematocrit > 30%
* Creatinine < 2.0 mg/dL
* Bilirubin < 2.0 mg/dL
* Albumin > 3.0 mg/dL
* No significant hepatic or renal dysfunction
* No other invasive cancer within the past 5 years
* No active infection or other active medical condition that could be eminently life threatening, including any of the following:

  * Active blood clotting
  * Bleeding diathesis
* No ongoing transfusion requirement
* No underlying cardiac disease associated with known myocardial dysfunction
* No unstable angina related to atherosclerotic cardiovascular disease
* No known autoimmune disease
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* Prior surgery, radiotherapy, chemotherapy, biological therapy (including sargramostim [GM-CSF]), or vaccine therapy allowed
* No concurrent anticancer therapy (e.g., hormone therapy for prostate or breast cancer)
* No concurrent digoxin or other medications for the treatment of heart failure
* No concurrent immunosuppressive therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Overall survival, progression-free survival, event-free survival, and failure-free survival
Frequency of immune response as measured by delayed-type hypersensitivity and serologic and cellular assays at baseline and during and after completion of study treatment
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Cancer Institute at Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

REFERENCES:
- [Derived] Nistor GI, Dillman RO. Cytokine network analysis of immune responses before and after autologous dendritic cell and tumor cell vaccine immunotherapies in a randomized trial. J Transl Med. 2020 Apr 21;18(1):176. doi: 10.1186/s12967-020-02328-6. PMID 32316978
- [Derived] Dillman RO, Cornforth AN, McClay EF, Depriest C. Patient-specific dendritic cell vaccines with autologous tumor antigens in 72 patients with metastatic melanoma. Melanoma Manag. 2019 May 31;6(2):MMT20. doi: 10.2217/mmt-2018-0010. PMID 31406564
- [Derived] Dillman RO, Cornforth AN, Depriest C, McClay EF, Amatruda TT, de Leon C, Ellis RE, Mayorga C, Carbonell D, Cubellis JM. Tumor stem cell antigens as consolidative active specific immunotherapy: a randomized phase II trial of dendritic cells versus tumor cells in patients with metastatic melanoma. J Immunother. 2012 Oct;35(8):641-9. doi: 10.1097/CJI.0b013e31826f79c8. PMID 22996370